CLINICAL TRIAL: NCT01165996
Title: A Proof of Concept Study of Non-DNA Damaging DNMT1 Depletion Therapy for Myelodysplastic Syndrome
Brief Title: Differentiation Therapy With Decitabine in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2908; NCI-2010-00135 (Other: NCI/CTRP); CASE2908 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-07-14; First posted 2010-07-20 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Myelodysplastic Syndromes; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Thrombocytopenia
Keywords: previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Thrombocytopenia | interventions — Flow Cytometry; DNA Methylation; Cytogenetic Analysis; Decitabine; Microarray Analysis; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I: decitabine (Experimental): INDUCTION PHASE: Patients receive decitabine subcutaneously (SQ) twice weekly for 4 weeks or thrice weekly until achieving bone marrow blasts < 5%. MAINTENANCE PHASE: Patients then receive decitabine SQ twice weekly for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: flow cytometry; Other: DNA methylation analysis; Other: cytogenetic analysis; Drug: decitabine; Genetic: microarray analysis; Genetic: gene expression analysis; Other: pharmacological study; Genetic: polymorphism analysis

INTERVENTIONS:
Other: flow cytometry — Correlative studies
Other: DNA methylation analysis — Correlative studies
Other: cytogenetic analysis — Correlative studies
Drug: decitabine — Given subcutaneously
  Other Names: 5-aza-dCyd; 5AZA; DAC; Dacogen; deoxyazacytidine; dezocitidine
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling
Genetic: gene expression analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Genetic: polymorphism analysis — Correlative studies

SUMMARY:
RATIONALE: Decitabine may help myelodysplastic cells become more like normal stem cells. PURPOSE: This clinical trial studies differentiation therapy with decitabine in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate that differentiation therapy with DNMT1 depleting but non-DNA damaging doses of decitabine is efficacious and can be administered weekly for > = 12 months. SECONDARY OBJECTIVES: I. Assess safety of the regimen.

II. Retrospectively compare study and standard regimen clinical responses. III. Assess the ability of a pharmacodynamic assay that measures DNMT1 depletion in peripheral blood white blood cells to predict clinical responses to decitabine.

IV. Assess PCR for aberrant methylation signature as an early marker of relapse. V. Identify biologic features of MDS that correlate with response to decitabine, thereby facilitating future patient selection.

VI. In cases of relapse or resistance, assess the role of the enzyme CDA in altering decitabine metabolism and preventing DNMT1 depletion.

OUTLINE:

INDUCTION PHASE: Patients receive decitabine subcutaneously (SC) twice weekly for 4 weeks or thrice weekly until achieving bone marrow blasts < 5%.

MAINTENANCE PHASE: Patients then receive decitabine SC twice weekly for up to 52 weeks in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* MDS classified by hematopathology review as WHO categories refractory anemia (RA) or refractory cytopenia with multi-lineage dysplasia (RCMD) or refractory anemia with ring sideroblasts (RARS) or refractory anemia with excess blasts (RAEB1 or RAEB2) or chronic myelo-monocytic leukemia (CMML1 or CMML2)
* Symptomatic anemia OR thrombocytopenia with a platelet count of < 100 x 10^9/L OR transfusion dependence for red-cells OR transfusion dependence for platelets OR absolute neutrophil count < 1 x 10^9/L

Exclusion

* MDS of the WHO sub-types RA or RCMD with sole 5q- abnormality on cytogenetics unless failed lenalidomide (Revlimid) therapy
* Previous treatment with decitabine
* Untreated erythropoietin deficiency defined as an erythropoietin level of < 200 IU/L and erythropoietin replacement therapy for < 8 weeks (erythropoietin deficiency until corrected)
* Uncontrolled infection
* Severe sepsis or septic shock
* Current pregnancy or breast feeding
* The patient is of childbearing age, and is unwilling to use contraception and has not had a tubal ligation, hysterectomy, or vasectomy , or their partner is also unwilling to use an acceptable method of contraception as determined by the investigator
* Not able to give informed consent
* Altered mental status or seizure disorder
* ALT > 300 IU; or albumin < 2.0 mg/dL
* Creatinine > 2.5 mg/dl and creatinine clearance < 60ml/min
* B12, folate, or iron deficient, until corrected
* NYHA class III/IV status
* ECOG performance status > 2
* HIV positive or history of seropositivity for HIV
* Transformation to acute leukemia ( >= 20% myelo-blasts in marrow aspirate)
* Any experimental agents other than the study drug decitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogen Saunthararajah, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Brenda Cooper, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Derived] Saunthararajah Y, Sekeres M, Advani A, Mahfouz R, Durkin L, Radivoyevitch T, Englehaupt R, Juersivich J, Cooper K, Husseinzadeh H, Przychodzen B, Rump M, Hobson S, Earl M, Sobecks R, Dean R, Reu F, Tiu R, Hamilton B, Copelan E, Lichtin A, Hsi E, Kalaycio M, Maciejewski J. Evaluation of noncytotoxic DNMT1-depleting therapy in patients with myelodysplastic syndromes. J Clin Invest. 2015 Mar 2;125(3):1043-55. doi: 10.1172/JCI78789. Epub 2015 Jan 26. PMID 25621498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from medical clinic between July 2010 and September 2011.
Groups:
- Arm I: Decitabine 0.2mg/kg: INDUCTION PHASE: Patients receive decitabine subcutaneously (SQ) twice weekly for 4 weeks or thrice weekly until achieving bone marrow blasts < 5%. MAINTENANCE PHASE: Patients then receive decitabine SQ twice weekly for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I: Decitabine 0.2mg/kg
Started | 25
Induction Phase | 25
Maintenance Phase | 23
Completed | 23
Not Completed | 2
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 25
Age, Customized [Number; unit: participants]
  40-49 years | 1
  50-59 years | 1
  60-69 years | 8
  70-79 years | 9
  80-89 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response as Defined by IWG (International Working Group) Criteria for Myelodysplasia
Description: Complete Response (CR) include less than 5% marrow blasts without evidence of dysplasia and normalization of peripheral blood counts, including a hemoglobin level of 110 g/L or more, a neutrophil count of 1.5 × 109/L or more, and a platelet count of 100 × 109/L or more. For PR, patients must demonstrate all CR criteria if abnormal before treatment except that marrow blasts should decrease by 50% or more compared with pretreatment levels, or patients may demonstrate a less-advanced MDS disease category than prior to treatment. Stable disease (SD) is defined by failure to achieve at least a partial response but no evidence of progression. Disease progression (DP) includes at least 50% decrease from maximum remission in granulocytes or platelets, reduction in hemoglobin by greater than or equal to 2g/dL, or transfusion dependence. Hematologic improvement (HI) includes hemoglobin increase by at least 1.5g/dL, reduction in transfusions, increase of platelets, increase of neutrophil count
Time Frame: Formal assessment at week 12 for study primary end-point (hematologic improvement).
Population: All patients enrolled and that received any treatment.
Measure: Number; unit: participants
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 25
participants
  Hematologic Improvement | 7
  Complete Remission | 4
  Partial Remission | 0
  Stable Disease | 9
  Disease Progression | 5

2. Secondary Outcome: Number of Patients That Experience > Grade 2 Non-hematologic Toxicity by National Cancer Institute (NCI)/Cancer Therapy Evaluation Program (CTEP) v4 Criteria
Description: Incidence of treatment-emergent adverse events (AEs) will be presented in tables that include causality, seriousness, severity/grade, and whether the AE resulted in death or discontinuation of treatment, Laboratory data will be summarized in tables that show changes from pre-treatment values and frequencies of abnormal values. Descriptive statistics will also be provided.
Time Frame: up to 12 months of treatment
Population: All patients that received treatment.
Measure: Number; unit: participants
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 25
participants | 16

3. Secondary Outcome: Cytogenetic Response as Per IWG Criteria
Description: Described as the number of patients with a major cytogenetic response (refers to disappearance of a cytogenetic abnormality) or a minor cytogenetic response (50% or more reduction of abnormal metaphases).
Time Frame: at 12 months
Population: Patients that had cytogenetic abnormalities at baseline and were evaluable with follow-up metaphase karyotyping.
Measure: Number; unit: participants
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 11
participants
  complete cytogenetic remission | 5
  partial cytogenetic remission | 2
  no cytogenetic remission | 4

4. Secondary Outcome: Proportion of Patients With Pharmacodynamic Evidence of Drug Effect.
Description: Evidence of pharmacodynamic effect will be correlated with clinical response criteria. The pharmacodynamic effect of treatment is defined as the number of participants that had depletion DNMT1 with minimal DNA damage and cytotoxicity.
Time Frame: 6 weeks after treatment
Population: All subjects that had treatment with DNMT1 depletion.
Measure: Number; unit: participants
Groups:
- Arm I: Decitabine 0.2mg/kg: INDUCTION PHASE: Patients receive decitabine subcutaneously (SQ) twice weekly for 4 weeks or thrice weekly until achieving bone marrow blasts < 5%. MAINTENANCE PHASE: Patients then receive decitabine SQ twice weekly for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  flow cytometry: Correlative studies
  DNA methylation analysis: Correlative studies
  cytogenetic analysis: Correlative studies
  decitabine: Given subcutaneously
  microarray analysis: Correlative studies
  gene expression analysis: Correlative studies
  pharmacological study: Correlative studies
  polymorphism analysis: Correlative studies
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 25
participants | 25

5. Secondary Outcome: Proportion of Patients With Bone Marrow Evidence of Cytotoxicity.
Description: Cytotoxicity is the ability to destroy cells. This will be measured by taking bone marrow samples and measuring the damage to cells. The level of cell destruction will be correlated with clinical response criteria.
Time Frame: 6 weeks after treatment
Population: Patients with chromosomal abnormalities which were evaluable for follow-up karyotyping
Measure: Number; unit: participants
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 11
participants
  Complete cytogenetic remission | 5
  Partial cytogenetic remission | 2

6. Secondary Outcome: Proportion of Patients With Bone Marrow Evidence of Terminal Differentiation Response to Therapy.
Description: Number of participants who, after therapy, had more of the differentiated types of blood (red cells, platelets, and white cells) compared to abnormal bone marrow cells than before therapy
Time Frame: 6 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 25
participants | 11

7. Secondary Outcome: Proportion of Patients With Particular Genetic Abnormalities Detected by Whole Exome Sequencing Correlation With Clinical Response
Description: Proportion of patients with particular genetic abnormalities, including DNA Methyltransferase 1 (DNMT1) depletion, detected by whole exome sequencing correlation with clinical response
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Arm I: Decitabine 0.2mg/kg
Number analyzed (Participants) | 25
participants | 4

ADVERSE EVENTS:
Time Frame: Data collected from on treatment to completion of treatment over a 1 year period.
Description: Only grade 3 and above AEs were collected and all submitted as SAEs.
Groups:
- Arm I: INDUCTION PHASE: Patients receive decitabine subcutaneously (SQ) twice weekly for 4 weeks or thrice weekly until achieving bone marrow blasts < 5%. MAINTENANCE PHASE: Patients then receive decitabine SQ twice weekly for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 15/25
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=25)
Acute Left Popliteal DVT (Vascular disorders) | 1 (1)
aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bacterial infection (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Death (General disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (17)
fever (General disorders) | 1 (1)
Furuncle on left groin area (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Left Sided Chest Pain (General disorders) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 2 (4)
Orthostasis (Vascular disorders) | 1 (2)
Orthostatic Hypotension (Vascular disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Tooth Extraction (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No